CLINICAL TRIAL: NCT02065297
Title: Quantitative and Functional Study of TH17 Lymphocytes in Horton's Disease (HD)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: AUDIA-SAMSON HORTON TH17
Record Dates: First submitted 2014-02-13; First posted 2014-02-19 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Horton's Disease; Infectious Disease; Neoplasia; Solid Tumor; Hemopathy
MeSH Terms: conditions — Giant Cell Arteritis; Communicable Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Horton's disease
  Interventions: Other: 2 to 3 blood samples (at inclusion, at 3 months and at 6 months in cases of relapse)
- Infectious disease
  Interventions: Other: 1 blood sample
- Neoplasia
  Interventions: Other: 1 blood sample
- Control
  Interventions: Other: 1 blood sample

INTERVENTIONS:
Other: 1 blood sample
  Groups: Control; Infectious disease; Neoplasia
Other: 2 to 3 blood samples (at inclusion, at 3 months and at 6 months in cases of relapse)
  Groups: Horton's disease

SUMMARY:
The aim of this open, controlled, multicentre biomedical research study is to identify new markers specifically associated with Horton's disease. This would make it possible to improve the diagnosis and management of this disease.

Participation consists in taking one or several blood samples depending on the group patients/controls.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Patients who have provided written informed consent
* Patients with national health insurance cover
* Age: 50 to 90 years

Patients with Horton' s disease :

* at the diagnosis, before any treatment
* or in remission
* or in relapse

Patients with an infectious disease :

* Bacteriologically or radiologically confirmed
* Presenting an inflammatory syndrome defined by :
* CRP ≥ 10 mg / L
* and Fibrinogen ≥ 4 g / L or ESR ≥ 30 mm at H1

Patients with neoplasia ( solid tumour or hemopathy ) :

* At the diagnosis, before treatment by chemotherapy
* Presenting an inflammatory syndrome defined by:
* CRP ≥ 10 mg / L
* and Fibrinogen ≥ 4 g / L or ESR ≥ 30 mm at H1

Controls :

These are healthy volunteers recruited among blood donators at Dijon CHU, voluntary hospital personnel ( nurses, doctors and secretaries ), patients at the EPHAD ( Champmaillot centre for geriatric patients ) and patients without infectious, inflammatory, or auto-immune disease ( CRP < 5mg / L ) or cancer recruited from the investigating departments of Dijon CHU. They will be matched for age and sex.

* Age: 18 - 90 years
* Patients with national health insurance cover
* who have provided written informed consent
* Absence of an inflammatory syndrome ( CRP < 5 mg / L )

Exclusion Criteria :

* Any patient who does not meet the inclusion criteria

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Horton' s disease Patients with an infectious disease Patients with neoplasia ( solid tumor or hemopathy ) Healthy controls
Sampling Method: Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2009-07-28 (Actual); Primary Completion 2016-01-07 (Actual)

PRIMARY OUTCOMES:
Quantification of specific cytokines of the Th17 immune response (IL-17 A and IL-23) in the serum | Up to 6 months
Quantification of LTh17 by flow cytometry | Up to 6 months
Measurement of the activation level of genes specifically involved in Th17 response using RT-PCR on frozen mRNA | Up to 6 months
Measure the ability of Treg to proliferate and to synthesize IL-17 in response to different antigenic stimulations | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de BESANCON, Besançon
  - CHU de DIJON, Dijon
  - CH de METZ, Metz